CLINICAL TRIAL: NCT01114893
Title: Travoprost Five Day Posology Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Matt Walker, PhD, Alcon Research, Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-09-075
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-05

CONDITIONS: Open-angle Glaucoma (OAG); Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Travoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- TRAVATAN (Active Comparator): TRAVATAN 0.004% once daily
  Interventions: Drug: Travoprost 0.004%
- Travoprost Vehicle (Placebo Comparator): Travoprost Vehicle
  Interventions: Drug: Travoprost Vehicle
- Travoprost Group A (Experimental): Travoprost Group A
  Interventions: Drug: Travoprost (Groups A, B and C)
- Travoprost Group B (Experimental): Travoprost Group B
  Interventions: Drug: Travoprost (Groups A, B and C)
- Travoprost Group C (Experimental): Travoprost Group C
  Interventions: Drug: Travoprost (Groups A, B and C)

INTERVENTIONS:
Drug: Travoprost 0.004% — 1 drop in each eye once daily for five days, and 1 drop vehicle in each eye 7 times daily for 5 days
  Arms: TRAVATAN
Drug: Travoprost Vehicle — 1 drop in each eye 8 times daily for 5 days
  Arms: Travoprost Vehicle
Drug: Travoprost (Groups A, B and C) — 1 drop in each eye 8 times daily for 5 days
  Arms: Travoprost Group A; Travoprost Group B; Travoprost Group C

SUMMARY:
The purpose of this study is to determine the safety and efficacy of three concentrations of travoprost ophthalmic solution (Groups A, B and C) administered eight times daily.

ELIGIBILITY:
Inclusion Criteria:

1. either sex and any race/ethnicity, ≥18 years old
2. diagnosed with open-angle glaucoma, and/or ocular hypertension
3. meets the following IOP entry criteria:

   * Mean IOP ≥ 24 millimeters mercury (mmHg) in at least 1 eye, with the same eye qualifying at 8 AM on both the Eligibility Visit (Day 0) and Day 1
   * Mean IOP ≤ 36 mmHg in both eyes at 8 AM and 8 PM at the Eligibility Visit (Day 0), and at 8 AM on Day 1
4. satisfies all informed consent requirements; able to read, sign and date the informed consent

Exclusion Criteria:

1. females of childbearing potential not meeting protocol conditions
2. angle grade less than Grade 2 in either eye
3. cup to disc ratio greater than 0.8 (horizontal or vertical measurement) in either eye
4. severe central visual field loss in either eye
5. any abnormality preventing reliable applanation tonometry in either eye
6. hypersensitivity to prostaglandin analogues or to any component of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center For Trial Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRAVATAN | Travoprost Vehicle | Travoprost Group A | Travoprost Group B | Travoprost Group C
Started | 14 | 14 | 14 | 13 | 12
Completed | 14 | 14 | 14 | 13 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRAVATAN | Travoprost Vehicle | Travoprost Group A | Travoprost Group B | Travoprost Group C | Total
Number analyzed (Participants) | 14 | 14 | 14 | 13 | 12 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 9 | 4 | 3 | 32
  >=65 years | 6 | 6 | 5 | 9 | 9 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 6 | 9 | 8 | 37
  Male | 7 | 7 | 8 | 4 | 4 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Intraocular Pressure (IOP) Change From Baseline at 8 AM on Day 5
Description: Outcome measure shows how each treatment reduced eye pressure at 8 AM on Day 5 compared to the eye pressure at 8 AM before the start of treatment
Time Frame: 5 days
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Travatan 0.004% QD | Travoprost Vehicle | Travoprost Group A | Travoprost Group B | Travoprost Group C
Number analyzed (Participants) | 14 | 14 | 14 | 13 | 12
mm Hg | -9.8 [-12.5 to -7.0] | -2.9 [-4.7 to -1.0] | -5.0 [-6.7 to -3.3] | -6.5 [-8.7 to -4.4] | -6.8 [-8.5 to -5.0]

2. Secondary Outcome: IOP Change From Baseline at 8 PM on Day 5
Description: Outcome measure shows how each treatment reducted eye pressure at 8 PM on Day 5 compared to the eye pressure at 8 PM before the start of treatment
Time Frame: 5 Days
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Travatan 0.004% QD | Travoprost Vehicle | Travoprost Group A | Travoprost Group B | Travoprost Group C
Number analyzed (Participants) | 14 | 14 | 14 | 13 | 12
mm Hg | -3.9 [-6.2 to -1.5] | -0.9 [-2.6 to 0.7] | -2.7 [-4.3 to -1.2] | -5.7 [-7.5 to -3.9] | -4.8 [-6.1 to -3.6]

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | TRAVATAN | Travoprost Vehicle | Travoprost Group A | Travoprost Group B | Travoprost Group C
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 8/14 | 2/14 | 5/14 | 8/13 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRAVATAN (N=14) | Travoprost Vehicle (N=14) | Travoprost Group A (N=14) | Travoprost Group B (N=13) | Travoprost Group C (N=12)
Eye Pruritus (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Ocular Hyperaemia (Eye disorders) | 4 (4) | 0 (0) | 5 (5) | 5 (5) | 5 (5)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Eye Irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign Body Sensation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal Staining (Eye disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Headache (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No